CLINICAL TRIAL: NCT07339683
Title: Influence of Cervical Stabilization Exercises on Neural Tissue Mechanosensitivity in Patients With Chronic Nonspecific Neck Pain
Acronym: NP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, nada ashraf mohamed zuhairy, principle investigator : nada ashraf mohamed zuhairy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005984
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Neck Pain
Keywords: cervical stabilization; tissue mechanosensitivity; neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: cervical and scapulothoracic stabilization exercises.
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical and scapulothoracic stabilization exercises. (Experimental): forty patients will receive cervical and scapulothoracic stabilization exercises plus traditional therapy three times a week for six weeks
  Interventions: Other: cervical and scapulothoracic stabilization exercises.; Other: traditional therapy
- traditional therapy (Active Comparator): forty patients will receive traditional therapy three times a week for six weeks
  Interventions: Other: traditional therapy

INTERVENTIONS:
Other: cervical and scapulothoracic stabilization exercises. — the patients will receive cervical and scapulothoracic stabilization exercises in the form of activation of deep cervical flexors in the first two weeks, followed by scapulothoracic muscles activation for the third and fourth weeks and finally group of exercises that emphasis on increasing difficulty and progress to quadruped and standing.
  Arms: cervical and scapulothoracic stabilization exercises.
Other: traditional therapy — the patients will receive traditional therapy in the form of ultrasound, hot pack, cervical extensors stretching and deep flexor strengthening

SUMMARY:
this study will be conducted to investigate the effect of cervical stabilization exercises on cervical pain intensity, upper limbs mechanosensitivity, cervicovertebral angle, and cervical proprioception in individuals with chronic nonspecific neck pain

DETAILED DESCRIPTION:
Neck pain is the sensation of discomfort in the neck area. Neck pain can result from disorders of any of the structures in the neck, including the cervical vertebrae and intervertebral discs, nerves, muscles, blood vessels, esophagus, larynx, trachea, lymphatic organs, thyroid gland, or parathyroid glands.Forward head posture (FHP) is one of the commonly recognized types of poor head posture in the sagittal plane in patients with neck pain. FHP has been defined as 'any alignment in which the external auditory meatus is positioned anterior to the plumb line through the shoulder joint, with a general prevalence of about 64% in both males and females.Several studies reported the effect of cervical stabilization exercises on pain, ROM and cranio-cervical angle in patients with chronic non-specific neck pain. No studies have been concerned with measuring mechanosensitivity as an indicator technique of the effect of different modalities on chronic non-specific neck pain. With the proposal of the cervical and scapulothoracic stabilization program for patients with chronic non-specific neck pain secondary to forward head posture deviations.

ELIGIBILITY:
Inclusion Criteria:

* participants with age range from 18 to 36 years and BMI from 25 to 30kg/m2 will be recruited
* Participants having neck pain symptoms provoked by neck postures, neck movement, or palpation of the cervical musculature, for 3 months
* Patients with a craniovertebral angle of less than 50º

Exclusion Criteria:

* History of previous injury of the neck.
* History of surgical intervention at the neck.
* History of inflammatory joint disease affecting facet joints
* participants with congenital disorders of the cervical spine.
* participants who received pain medication or physical therapy for their neck pain during the last 3 months.

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
mechanosensitivity of upper limb nerves | up to 6 weeks
  A handheld algometer will be used to assess mechanosensitivity. To apply this test test, specific points on the peripheral nerve trunks of the tested upper limb nerves will be identified through manual palpation, being easily accessible by the probe of the algometer and as they are commonly used sites of peripheral nerves' palpation with moderate inter-tester reliability. The supine lying posture will be assumed to test median and ulnar nerves, while sitting posture will be the choice for radial nerve. Median nerve will be located and tested in the antebrachial fossa just medial to the biceps brachii tendon. Ulnar will be tested in the cubital tunnel between humeral medial epicondyle and olecranon process, with the arm in 90º shoulder abduction as well as external rotation, and elbow flexion. Radial nerve palpation point lies between the middle and lower thirds of the humerus.

SECONDARY OUTCOMES:
craniovertebral angle | up to 6 weeks
  craniovertebral angle will be assessed by Kinovia software. Forward head posture will be determined when the craniovertebral angle is below 50 degrees (normal value).
pain intensity | up to six weeks
  Visual analogue scale is the most commonly used method for assessing pain intensity. The left most value on the 10-cm horizontal line used for visual analogue scale indicates a painless condition, which is represented by 0. The rightmost value is 10, which represents extreme pain. The subjects will be in a relaxed position then will give them the appendix which contains VAS and rate their feelings of pain on the line by themselves, thereby quantifying the pain
cervical joint position error (cervical proprioception) | up to six weeks
  To evaluate the joint position error , the examiner will hold the subject's head and moving slowly to the target head position, which is 50% of the maximum CROM and hold there for a period of 3 s. The subjects then memorized that target position and then the examiner slowly brought the subject's head back to the neutral position. The subjects then will be advised to reach the target position actively by moving the head and when subject reached the target position the reposition accuracy error will determine in degrees. The examiner will evaluate JPE tests in sagittal (flexion, extension) and transverse plane (right and left rotation) directions. Each direction of JPE testing will be performed three times and the mean error of these trials will be used in the analysis